CLINICAL TRIAL: NCT04079504
Title: Comparison of Postoperative Pain After Hernial Sac Ligation Versus Non-ligation in Inguinal Hernioplasty.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syed Ali Haider, Assistant Professor of Surgery, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-1286/DUHS
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Inguinal Hernia, Indirect; Postoperative Pain
Keywords: Indirect inguinal hernia; Ligation of sac; Postoperative pain
MeSH Terms: conditions — Hernia, Inguinal; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ligation (Active Comparator): Ligation of indirect inguinal hernia sac in inguinal hernioplasty patients
  Interventions: Procedure: Ligation of indirect hernia sac
- Non-ligation (Experimental): Non-Ligation of Indirect inguinal hernia sac/ simple inversion/reduction of indirect inguinal hernia sac in inguinal hernioplasty patients
  Interventions: Procedure: Non-ligation of Indirect Inguinal hernia sac

INTERVENTIONS:
Procedure: Ligation of indirect hernia sac — Indirect inguinal hernia sac will be separated from the spermatic cord and contents of the sac will be reduced before ligating it at the deep inguinal ring.
  Other Names: Prolene Mesh Placement
  Arms: Ligation
Procedure: Non-ligation of Indirect Inguinal hernia sac — the indirect inguinal hernia sac will be separated from the spermatic cord and reduced/inverted in to the peritoneal cavity through the deep inguinal ring along with its contents.
  Other Names: Prolene Mesh placement
  Arms: Non-ligation

SUMMARY:
This study is intends to compare mean postoperative pain scores for 48-hours in patients undergoing Inguinal hernioplasty with and without hernia sac ligation in Department of Surgery, Dow University of Health Sciences & Dr. Ruth K. M. Pfau Civil Hospital Karachi.Half of the patients undergoing inguinal hernioplasty will have their indirect inguinal sacs ligated whereas other half will have non-ligation and inversion of sac.

DETAILED DESCRIPTION:
Amongst general surgical operations done in elective theaters, Hernioplasty is one of the most common. In the current era of new and developing maneuvers of inguinal hernia repairs, the conventional anterior, tension-free approach is considered a daycare method with minimal morbidities. However, mild to medium early postoperative pain is frequent with reported incidence of 21.6% in literature.

The reasons of postoperative pain after hernia repair are multifactorial. Delikoukos et al mentioned that ilioinguinal nerve entrapment or mesh fixation in the periosteum of the pubic tubercle are major etiological factors in the occurrence of postoperative pain. Later studies highlighted that these factors are major culprits in chronic neuralgias with inconsistent involvement in early postoperative pain after mesh repair.This necessitated the exploration of other offenders causing early postoperative pain. In this context, surgeons focused on the role of hernial sac ligation in mesh repairs of indirect inguinal hernias. The notion behind this operative technique is the generation of pain as a consequence of highly pain sensitive parietal peritoneum trauma during ligation and division of hernia sac, the fact which was highlighted by Schulman et al nearly two decades ago. Despite this imperative reason, there is a noteworthy gap on this aspect of early pain with studies still addressing the chronic pain after mesh repair of inguinal hernias. A research reports that frequency of early postoperative pain at day one was significantly higher in 'hernial sac high ligation group' as compared to 'hernial sac non-ligation group' (mean postoperative pain on VAS; 3.5±1.5, and 2.3±1.2 respectively, p<0.05), yet other studies report no significant difference in pain when evaluating different operative techniques.However further studies are needed to establish omission of hernia sac ligation as part of the standard procedure.

Early postoperative pain not only results in delayed recovery and return to normal activity but also adds to the financial constraints of patient and health system.Therefore, the aim of this study is to compare the early postoperative pain after hernia sac ligation as compared to non-ligation in order to establish a definitive role of these operative techniques in the development of early postoperative pain after mesh repair of inguinal hernia so the superior of the two techniques will be employed subsequently.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥15 years of age, of either gender having Incomplete indirect inguinal hernia with or without direct concurrent hernia as mentioned in operational definition.

Exclusion Criteria:

* Complete inguinal hernias.
* Patients having obstructed and/or strangulated inguinal hernia.
* Recurrent inguinal hernias.
* patients with ipsilateral synchronous inguinoscrotal pathologies e.g. hydrocele, testicular malignancy

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
Mean Postoperative pain | up to 48 hours
  Pain scores on visual Analogue scale (0-10) at 12,24,36,48 hours after surgery, Mean will be calculated

SECONDARY OUTCOMES:
Duration of Surgery | Baseline(at the time of surgery)
  Duration of operations in both arms will be recorded and mean will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Syed A Haider, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences & Dr. Ruth K. M. Pfau Civil Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Delikoukos S, Lavant L, Hlias G, Palogos K, Gikas D. The role of hernia sac ligation in postoperative pain in patients with elective tension-free indirect inguinal hernia repair: a prospective randomized study. Hernia. 2007 Oct;11(5):425-8. doi: 10.1007/s10029-007-0249-9. Epub 2007 Jun 27. PMID 17594052
- [Background] Mohta A, Jain N, Irniraya KP, Saluja SS, Sharma S, Gupta A. Non-ligation of the hernial sac during herniotomy: a prospective study. Pediatr Surg Int. 2003 Aug;19(6):451-2. doi: 10.1007/s00383-002-0940-y. Epub 2003 May 28. PMID 12774253
- [Background] Shulman AG, Amid PK, Lichtenstein IL. Ligation of hernial sac. A needless step in adult hernioplasty. Int Surg. 1993 Apr-Jun;78(2):152-3. PMID 8354615